CLINICAL TRIAL: NCT06340685
Title: An Open Label, Exploratory, Proof-of Concept Study of Triheptanoin as Treatment for Patients With Primary-Specific Pyruvate Dehydrogenase Complex (PDC) Deficiency
Brief Title: Triheptanoin for Children With Primary-Specific Pyruvate Dehydrogenase Complex (PDC) Deficiency
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jirair Krikor Bedoyan (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Jirair Krikor Bedoyan, Associate Professor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23050042; UX007-IST236 (Other Grant/Funding Number: Ultragenyx Pharmaceutical Inc.)
Record Dates: First submitted 2024-03-22; First posted 2024-04-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Pyruvate Dehydrogenase Complex Deficiency
Keywords: Pyruvate Dehydrogenase Complex Deficiency
MeSH Terms: conditions — Pyruvate Dehydrogenase Complex Deficiency Disease | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Triheptanoin (Experimental): Open label study
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — Open-label design with doses of triheptanoin up to 4.0 gm/kg triheptanoin
  Other Names: Dojolvi

SUMMARY:
This is a medical research study to test a medication in patients with a disease called Pyruvate Dehydrogenase Complex (PDC) Deficiency. The medication is triheptanoin, which is currently FDA approved for the treatment of Long-Chain Fatty Acid Oxidation Disorders. Previous research suggests that triheptanoin may also be effective in the treatment PDC Deficiency. This study will investigate the safety and efficacy (how well it works) of triheptanoin in patients with PDC Deficiency.

DETAILED DESCRIPTION:
Participation in the study will require the patient to participate in up to 10 visits over a two-year period. Five of those visits must be done at the UPMC Children's Hospital of Pittsburgh (CHP). Other visits can take place at CHP or remotely. All of these visits will include blood draws.

Triheptanoin will be added to the patients' diet and administered at least 4 times per day. The target dose will be 1.2-3.9 g of triheptanoin per kg body weight with a max goal dose of about 4 g/kg per day.

The triheptanoin will be provided to the patients at no cost. All other costs will be billed to the patients' insurance.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1 year to <18 years of age
2. Subjects with PDCD would need to have a metabolic physician following their clinical care needs prior to their enrollment in the study
3. Diagnosis of PDCD by molecular genetic confirmation of PDHA1, PDHB, DLAT, PDHX, or PDP1 mutation
4. Not pregnant or lactating
5. Parental permission and assent of minor and willingness to comply with study procedures
6. Not participating in any interventional treatment clinical trials
7. Not a recipient of gene therapy, organ transplant, or bone-marrow transplantation
8. If currently on any investigational drugs or therapies, must complete a 30-day washout period prior to Intake & Dosing (Day 1).
9. Negative pregnancy test for all female patients of childbearing age. Individuals of childbearing potential must agree to use a highly effective method of contraception, and males must agree not to father a child or donate sperm. True abstinence for the duration of the study will also be accepted.
10. Subjects are following some form or type of ketogenic diet at the time of the screening visit.

Exclusion Criteria:

1. Diagnosis of medium-chain acyl-CoA dehydrogenase (MCAD)
2. Use of alcohol or drugs of abuse
3. Evidence of liver disease as defined by elevations of AST or ALT >2x ULN in the past 6 months
4. Pregnant, breastfeeding, or lactating females
5. On any investigational product research study (and not completed the required 30-day washout period prior to Intake & Dosing) or recipient of gene therapy or organ or bone-marrow transplantation

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who report side-effects related to gastrointestinal (GI) distress | 24 months
Normalization of biochemical markers of disease (lactate) | 24 months
  Change in lactate levels, comparing results from before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in mmol/L
Normalization of biochemical markers of disease (pyruvate) | 24 months
  Change in pyruvate levels, comparing results from before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in mg/dl
Normalization of biochemical markers of disease (β-hydroxybutyrate level) | 24 months
  Change in β-hydroxybutyrate levels, comparing results from before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in mmol/L
Normalization of biochemical markers of disease (Alanine/Leucine ratio) | 24 months
  Change in Alanine/Leucine ratios, comparing results from before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in μmol/L
Normalization of biochemical markers of disease (Alanine/Lysine ratio) | 24 months
  Change in Alanine/Lysine ratios, comparing results from before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in μmol/L
Normalization of biochemical markers of disease (Alanine/Proline ratio) | 24 months
  Change in Alanine/Proline ratios, comparing results from before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in μmol/L
More efficacious seizure control | 24 months
  Measured by a reduction or alteration of home antiepileptics use, from before and after triheptanoin is initiated
More efficacious metabolic control | 24 months
  Measured by a reduction in episodes of metabolic decompensation, from before and after triheptanoin is initiated
More efficacious disease control | 24 months
  Measured by a reduction in the frequency of disease related hospitalizations, from before and after triheptanoin is initiated

SECONDARY OUTCOMES:
Improved quality of life | 24 months
  Measured by a change in scores on the PedsQL, from before and after trihepatnoin is initiated
Improved long-term maintenance and tolerance of diet | 24 months
  Measured by parental report of diet maintenance and tolerance, from before and after triheptanoin is initiated
Improved quality of life | 24 months
  Measured by a change in scores on the MetabQoL, from before and after trihepatnoin is initiated

CONTACTS AND LOCATIONS:
Overall Officials: Jirair Bedoyan, MD, PhD, Principal Investigator — UPMC Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No